CLINICAL TRIAL: NCT06281028
Title: SOLACEA-H vs HYDROLINK-NVU for Haemodialysis Sessions in Extracorporeal Circulation Heparin-sparing Situations
Brief Title: SOLACEA-H in Heparin-sparing Haemodialysis
Acronym: SOLHEPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A02280-45
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Dialysis Membrane Reaction

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A : SOLACEA-H/HYDROLINK-NVU (Other): The dialysis sessions will take place in the following order :
  Wash - SOLACEA-H dialysis - Wash - HYDROLINK-NVU dialysis
  Interventions: Device: SOLACEA-H/HYDROLINK-NVU
- B : HYDROLINK-NVU/SOLACEA-H (Other): The dialysis sessions will take place in the following order :
  Wash - HYDROLINK-NVU dialysis - Wash - SOLACEA-H dialysis
  Interventions: Device: HYDROLINK-NVU/SOLACEA-H

INTERVENTIONS:
Device: SOLACEA-H/HYDROLINK-NVU — Patients will receive 6 sessions of washout treatment, followed by a gradual tapering phase (4 sessions maximum) during which the anticoagulant will be reduced from the normal dose to the minimum effective dose (which may be zero) and maintained for a minimum of 2 sessions on the SOLACEA-H, followed by 6 washout sessions, then again a gradual reduction phase (4 sessions maximum) during which the anticoagulant will be reduced from the normal dose to the minimum effective dose (which may be zero) and maintained for a minimum of 2 sessions on the HYDROLINK-NVU.
  Arms: A : SOLACEA-H/HYDROLINK-NVU
Device: HYDROLINK-NVU/SOLACEA-H — Patients will receive 6 sessions of washout treatment, followed by a gradual tapering phase (4 sessions maximum) during which the anticoagulant will be reduced from the normal dose to the minimum effective dose (which may be zero) and maintained for a minimum of 2 sessions on the HYDROLINK-NVU, followed by 6 washout sessions, then again a gradual reduction phase (4 sessions maximum) during which the anticoagulant will be reduced from the normal dose to the minimum effective dose (which may be zero) and maintained for a minimum of 2 sessions on the SOLACEA-H.
  Arms: B : HYDROLINK-NVU/SOLACEA-H

SUMMARY:
The aim of the study is to evaluate the efficacy of the SOLACEA-H dialyser, particularly in patients at high risk of haemorrhage, during post-dilution haemodiafiltration sessions with complete or partial heparin sparing. It will be compared with another dialyser (HYDROLINK-NVU)

DETAILED DESCRIPTION:
This is a randomised, crossover, open-label, prospective, multicentre post-marketing clinical follow-up study comparing two medical devices used (SOLACEA-H dialyser vs HYDROLINK-NVU dialyser) for their intended purpose.

Each patient will be followed for approximately 2 months, depending on the number of sessions in the anticoagulant reduction phase.

Patients will be offered the study by the investigator during a dialysis session as part of routine practice. If the patient accepts and signs the informed consent form, he or she will receive a succession of dialysis sessions including first the SOLACEA-H then the HYDROLINK-NVU membrane, or vice versa, depending on randomisation.

ELIGIBILITY:
Inclusion Criteria:

* On haemodialysis for at least 3 months
* Dialysis in a haemodialysis department of the Ramsay-Santé group
* No active infection
* Medically stable
* Blood flow ≥ 300 ml/min
* Haemoglobin level stable and within recommended norms for a dialysis patient, id est > 10g/dl
* Bipunction
* No known allergy to SOLACEA H or HYDROLINK-NVU
* Willingness to comply with study procedures for the duration of the study
* For women of childbearing age: effective contraception, or absence of active pregnancy (negative pregnancy test)
* Member or beneficiary of a social security scheme
* Patient having been informed and having signed an informed consent form

Exclusion Criteria:

* Patient on oral anticoagulants for the duration of the study
* Patient on dialysate for the duration of the study
* Patient Medically unstable or fragile
* Severe hepatic impairment
* Patient hospitalised without consent
* Concurrent participation in another clinical study
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, breast-feeding or parturient women
* Patient unable to receive heparin
* Known allergy to latex or phthalates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
SOLACEA-H vs HYDROLINK-NVU efficacy | 2 month
  The primary endpoint is dialysis time, as a marker of a complete and successful dialysis session. This criterion will make it possible to evaluate the effectiveness of a dialysis treatment with SOLACEA-H, complete without total coagulation of the circuit with little or no anticoagulant , with a similar or lesser quantity than that used for the current treatment with HYDROLINK-NVU.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé La Louvière, Lille, France